CLINICAL TRIAL: NCT01742351
Title: Internet-based Cognitive Behaviour Therapy for Persons Diagnosed With Bipolar II - a Pilot Study
Brief Title: Internet-based Cognitive Behaviour Therapy (CBT) for Persons Diagnosed With Bipolar II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro County Council (Other Government)
Collaborators: School of Law, Psychology and Social Work, Örebro University (Unknown)
Responsible Party: Principal Investigator, Fredrik Holländare, Psychologist, PhD, Örebro County Council
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 39:2012
Record Dates: First submitted 2012-11-16; First posted 2012-12-05 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Bipolar Disorder, Type II
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Guided internet-based cognitive behavior therapy (CBT) (Experimental)
  Interventions: Behavioral: Guided internet-based cognitive behavior therapy

INTERVENTIONS:
Behavioral: Guided internet-based cognitive behavior therapy

SUMMARY:
The aim of the study is to test the feasibility and acceptability of internet-based Cognitive Behaviour Therapy (CBT) for persons diagnosed with bipolar disorder, type II. The idea is to treat residual depressive symptoms as well as using psychoeducation to improve their prognosis. Each participant will have a personal therapist that will provide guidance and support throughout the treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of bipolar disorder type II
* Mild to moderate depressive symptoms
* 18 years of age
* Stable medication with a mood stabiliser
* Access to the internet

Exclusion Criteria:

* Diagnosis of psychosis
* Having received psychiatric in-patient care during the past year
* Ongoing psychotherapy
* Previous manic episode
* Previous suicide attempt
* Previous parasuicidal behavior documented in patient record (e.g. self-injury)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in score on the Montgomery-Åsberg Depression Rating Scale - Self rated (MADRS-S) between baseline and post treatment | 9 weeks
  A nine item questionnaire of depressive symptoms

SECONDARY OUTCOMES:
Change in the score on the Affective Self Rating Scale (AS-18-M) between baseline and post treatment | 9 weeks
  A nine item subscale of the AS-18 measuring symptoms of mania/hypomania.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Holländare, PhD, Principal Investigator — School of Health and Medical Science, Psychiatric Research Centre
Locations (1):
- Psychiatric Research Centre, Örebro, Sweden

REFERENCES:
- [Derived] Hollandare F, Eriksson A, Lovgren L, Humble MB, Boersma K. Internet-Based Cognitive Behavioral Therapy for Residual Symptoms in Bipolar Disorder Type II: A Single-Subject Design Pilot Study. JMIR Res Protoc. 2015 Apr 23;4(2):e44. doi: 10.2196/resprot.3910. PMID 25908235